CLINICAL TRIAL: NCT06224088
Title: Neuro-cognitive Function 1 Year Post ICU Discharge Among VV ECMO Survivors: a Prospective Observational Study
Brief Title: Neuro-cognitive Function 1 Year Post ICU Discharge Among VV ECMO Survivors
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: 0015-24-MMC
Record Dates: First submitted 2024-01-15; First posted 2024-01-25 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Neurocognitive Dysfunction
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: VV ECMO — treatment with VV ECMO in the ICU

SUMMARY:
In the past three years, in the general intensive care unit in Meir medical center, 25 patients were treated with ECMO, of which two patients were treated with VA ECMO and the rest with VV ECMO. 70% of the patients survived to hospital discharge.

ECMO is indicated as a rescue therapy for patients in critical condition suffering from severe cardiac and/or respiratory failure that does not respond to conservative treatment. It can be used as a bridge to recovery or to heart/lung transplantation. ECMO was introduced in the late seventies of the pervious century. Between the years 2006-2011, partly due to the outbreak of the flu epidemic (H1N1), a 433% increase was observed in the use of ECMO worldwide in adults. In light of the outbreak of the Covid-19 epidemic in recent years, another significant increase has been observed.

There are short-term and long-term complications of ECMO. Short-term complications include bleeding, thrombosis, hemolysis, HIT, renal and neurological injuries, associated infections, and technical-mechanical problems. Long-term complications include significant physical and psychological consequences that may adversely affect the patient's daily function, especially executive function.

ELIGIBILITY:
Inclusion Criteria: All patients treated with VV ECMO who survived to hospital discharge between 2021-2023 -

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with VV ECMO who survived to hospital discharge between 2021-2023
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Neurocognitive function in ECMO survivors as measured by SF-36 questionnaire | one year after hospital discharge
  Neurocognitive function in ECMO survivors one year after hospital discharge as measured by SF-36 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: Undecided